CLINICAL TRIAL: NCT02408848
Title: Three Dimensional Echocardiography in Congenital Cardiac Surgery
Brief Title: The Value of Three Dimensional Echocardiography in Congenital Cardiac Surgery
Status: Terminated | Type: Observational
Why Stopped: No three dimensional transthoracic echo available currently
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Mona Momeni, MD, PhD, Chef de Clinique associée, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: 2015/06JAN/006
Record Dates: First submitted 2015-03-18; First posted 2015-04-06 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Observational — This is an observational study. There is no intervention.

SUMMARY:
There are few studies evaluating the value of 3D echocardiography in children undergoing congenital cardiac surgery. The aim of this observational study is to describe common and uncommon congenital malformations with the help of 3D echo and compare the findings and the measurements with those obtained with conventional 2D echo.

ELIGIBILITY:
Inclusion Criteria:

* All children requiring general anesthesia for congenital heart surgery and in whom informed parental consent has been obtained

Exclusion Criteria:

* Children with congenital heart disease who do not require heart surgery

Ages: 5 Hours to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing congenital cardiac surgery with or without cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
correlate three dimensional measurements with two dimensional measurements | 1 month
  correlation of two dimensional transthoracic echo with three dimensional transthoracic echo

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium